CLINICAL TRIAL: NCT03523377
Title: Overnight Fasting After Completion of Therapy: The OnFACT Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-199
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Childhood Cancer Survivors
Keywords: Fasting; 18-199
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Intervention Model Description: The OnFACT study is a pilot randomized controlled trial of prolonged overnight fasting among adult survivors of childhood cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prolonged overnight fasting (Experimental): Participants randomized to the fasting arm will be instructed on how to use the SMS texting app to indicate the beginning and end of the nightly fast. In the first 2-4 weeks following the first overnight fast, intervention participants will complete three phone calls with study staff trained in motivational interviewing. These calls will be used to reinforce the prolonged overnight fasting instructions, identify barriers to prolonged overnight fasting, and support successes where they have occurred.
  Interventions: Other: prolonged overnight fasting
- usual care (Active Comparator): Participants randomized to the usual care arm will be instructed to eat a heart-healthy diet and exercise for at least 30 minutes five days a week, which is usual counseling in our clinics.
  Interventions: Other: usual care

INTERVENTIONS:
Other: prolonged overnight fasting — Three phone calls using motivational interviewing, support via SMS text.
  Arms: prolonged overnight fasting
Other: usual care — Eat a heart-healthy diet and exercise for at least 30 minutes five days a week
  Arms: usual care

SUMMARY:
The purpose of this study is to test whether regularly not eating for at least 14 hours overnight ("intermittent fasting") is feasible and can improve blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index is ≥ 18.5 kg/m^2
* History of treatment for cancer or related illness diagnosed at ≤ 25 years old
* Off cytotoxic therapy for primary cancer ≥ 2 years
* Not receiving cytotoxic therapy (chemotherapy, external beam radiation therapy) at the time of study enrollment
* History of radiation to the chest, abdomen or total body
* Current age ≥18 years
* English-speaking
* Personal phone with SMS text messaging capability
* Willingness to wear an mHealth device, such as a FitBit, for two 7-day periods
* Able to perform all study requirements

Exclusion Criteria:

* Use of any antidiabetic, weight loss, or appetite control medication
* Use of any other medication that could impact dietary intake, such as prednisone
* Currently fasts 12 hours or more by self-report
* Unable to fast due to medical reason such as pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Participation completion | 6 months
  Proportion of registered participants who successfully complete the 6-month intervention

SECONDARY OUTCOMES:
measure of glucose metabolism | 6 months
  Assess the effect of prolonged overnight fasting on glucose metabolism, measured by glycosylated hemoglobin (HbA1c).

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Friedman, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm